CLINICAL TRIAL: NCT03999398
Title: Short and Long-term Results of PCI in no Touch Vein-graft:a Comparison With the Standard One.
Brief Title: Short and Long-term Results of PCI in no Touch Vein-graft.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Region Örebro County (Other)
Collaborators: Karlstad Central Hospital (Other)
Responsible Party: Principal Investigator, Gabriele Ferrari, Medical Doctor, Region Örebro County
Other Study IDs: OLL-242381
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Percutaneous Coronary Intervention; Saphenous Vein; Coronary Artery Bypass
Keywords: Saphenous Vein; No-touch; Percutaneous Coronary Intervention
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No-touch: Participants that operated at the time of the coronary artery bypass grafting with a "no-touch" venous graft.
  Interventions: Procedure: Percutaneous coronary intervention (PCI)
- Conventional: Participants that operated at the time of the coronary artery bypass grafting with a "conventional" venous graft.
  Interventions: Procedure: Percutaneous coronary intervention (PCI)

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI) — Participants are treated with a PCI and stent implantation in a venous graft (previously implanted during the CABG operation)
  Other Names: Previously: coronary artery bypass grafting (CABG)

SUMMARY:
Coronary artery disease is one of the biggest health issue worldwide.The treatment, in a large part of the patients, implicates a so called bypass-operation, that consists in to connect new vascular conduits (grafts) beyond the narrowed coronary vessels to improve the blood supply to the heart. One of the graft that is commonly used is the saphenous vein from the leg. The disadvantage of the saphenous vein graft is the predisposition to early obstruction. The international literature shows the following grades of occlusion: 15% in the first year and 40% after 10 year.

At the Cardio-Thoracic Clinic of the University hospital of Örebro has been developed a new method to harvest the saphenous vein together with the surrounding fat-tissue. This technique, called no-touch technique, has the advantage to reduce the damages to the vein during the harvesting, showing a substantially reduced risk for future occlusion (5% after 18 months and 10% after 8,5 years).

The aim of the PhD project is to evaluate the results of the no-touch technique in compare to the conventional technique for the venous graft harvesting. The focus of the study is to analyse all the operated patients in our clinic who underwent a post-operative coronary angiography do to angina pectoris (heart pain). All the patients who received a stent during the post-operative angiography will be analysed in detail and one will compare the occlusion grade and the rate of major adverse cardiac events (MACE).

This study is the first and the only one in the world that will examine the long-term results of the no-touch technique in particular after the stenting of the venous graft.

DETAILED DESCRIPTION:
The study is a observational retrospective with registered-based data. The register used is Swedeheart which is the national Swedish intervention-related quality register for cardiological interventions (such as percutaneous coronary intervention (PCI)) and cardiac surgical procedures that are performed every year in Sweden.

After the approval of the Regional ethical review board in Uppsala (Sweden), one could review all the subjects that received a PCI in a venous graft between January the 1st, 2006 and June the 30th, 2020 either at the Angiographic unit of the University Hospital of Orebro or at the Angiographic unit of the Hospital of Karlstad. All the participants has been previously operated at the Cardiothoracic department of the University hospital of Orebro with a coronary artery bypass grafting (CABG) procedure, with one type of vein graft (no-touch) or the other (standard) All the relevant data for the study that are missed in the quality register, are extrapolated by the clinical registers of the two hospital involved (Orebro and Karlstad).

Once finished the data extraction and review, the data will be statistically analysed in term of short and long term results; and an advanced comparison between the two different type of venous graft involved. This is to show if there is a significant difference between the two techniques also after a PCI procedure (already proven clinical different between the two technique in favour of the no-touch one by numerous studies).

Moreover an assessment of the patients´ quality of life in the two different studies will be performed with the use of Health related quality of life surveys (RAND-36); even a health economics analysis will be preformed (QALY).

ELIGIBILITY:
Inclusion Criteria:

* Participants previously operated with a coronary artery bypass grafting at the Cardiothoracic department of the University hospital of Orebro
* Participants that underwent a percutaneous coronary intervention in a venous graft

Exclusion Criteria:

* percutaneous coronary intervention within 30 days from the primary operation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the subjects that previously were operated with a coronary artery bypass grafting at the Cardiothoracic department of the University hospital of Orebro (from the 1992 until 30th June 2020) and that underwent a percutaneous coronary intervention in a venous graft between January the 1st, 2006 and June the 30th, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-02 (Estimated)

PRIMARY OUTCOMES:
Rate of In-stent restenosis | after the percutaneous coronary intervention (until December the 01st 2020)
  stenosis or occlusion of the stent implanted during the percutaneous coronary intervention procedurerevascularisation)

SECONDARY OUTCOMES:
Rate of Major adverse cardiac event (MACE) | after the percutaneous coronary intervention (until December the 01st 2020)
  adverse cardiac event (mortality (cardiac) + myocardial infarction + target vessel
Quality of life (RAND-36) | after the percutaneous coronary intervention, through study completion, an average of 5 years
  health related quality of life surveys assessment; reporting a score on a scale,the minimum value is 0 and the maximum value is 100; higher scores mean a better outcome
QALY (quality-adjusted life-year) | after the percutaneous coronary intervention, through study completion, an average of 5 years
  health economics analysis

OTHER OUTCOMES:
Rate of Mortality | after the percutaneous coronary intervention (until December the 01st 2020)
  overall mortality after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Ferrari, MD, Principal Investigator — Region Örebro län
Locations (1):
- Kärl-Thoraxkliniken; University Hospital of Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: All the individual data that can be shared according the Regional ethical review board rules. Those data will be share a specific upon request in order to contribute to other researchers own works (that want to compare their results with ours) or in case of meta-analysis.

REFERENCES:
- [Background] Souza D. A new no-touch preparation technique. Technical notes. Scand J Thorac Cardiovasc Surg. 1996;30(1):41-4. doi: 10.3109/14017439609107239. No abstract available. PMID 8727856
- [Background] Souza DS, Dashwood MR, Tsui JC, Filbey D, Bodin L, Johansson B, Borowiec J. Improved patency in vein grafts harvested with surrounding tissue: results of a randomized study using three harvesting techniques. Ann Thorac Surg. 2002 Apr;73(4):1189-95. doi: 10.1016/s0003-4975(02)03425-2. PMID 11996262
- [Background] Souza DS, Johansson B, Bojo L, Karlsson R, Geijer H, Filbey D, Bodin L, Arbeus M, Dashwood MR. Harvesting the saphenous vein with surrounding tissue for CABG provides long-term graft patency comparable to the left internal thoracic artery: results of a randomized longitudinal trial. J Thorac Cardiovasc Surg. 2006 Aug;132(2):373-8. doi: 10.1016/j.jtcvs.2006.04.002. PMID 16872965
- [Background] Samano N, Bodin L, Karlsson J, Geijer H, Arbeus M, Souza D. Graft patency is associated with higher health-related quality of life after coronary artery bypass surgery. Interact Cardiovasc Thorac Surg. 2017 Mar 1;24(3):388-394. doi: 10.1093/icvts/ivw372. PMID 28040753
- [Background] Samano N, Geijer H, Liden M, Fremes S, Bodin L, Souza D. The no-touch saphenous vein for coronary artery bypass grafting maintains a patency, after 16 years, comparable to the left internal thoracic artery: A randomized trial. J Thorac Cardiovasc Surg. 2015 Oct;150(4):880-8. doi: 10.1016/j.jtcvs.2015.07.027. Epub 2015 Jul 15. PMID 26282605
- [Background] Bourassa MG. Fate of venous grafts: the past, the present and the future. J Am Coll Cardiol. 1991 Apr;17(5):1081-3. doi: 10.1016/0735-1097(91)90835-w. No abstract available. PMID 2007707
- [Background] Campeau L, Enjalbert M, Lesperance J, Bourassa MG, Kwiterovich P Jr, Wacholder S, Sniderman A. The relation of risk factors to the development of atherosclerosis in saphenous-vein bypass grafts and the progression of disease in the native circulation. A study 10 years after aortocoronary bypass surgery. N Engl J Med. 1984 Nov 22;311(21):1329-32. doi: 10.1056/NEJM198411223112101. PMID 6333635
- [Background] Fitzgibbon GM, Kafka HP, Leach AJ, Keon WJ, Hooper GD, Burton JR. Coronary bypass graft fate and patient outcome: angiographic follow-up of 5,065 grafts related to survival and reoperation in 1,388 patients during 25 years. J Am Coll Cardiol. 1996 Sep;28(3):616-26. doi: 10.1016/0735-1097(96)00206-9. PMID 8772748
- [Background] Hindnavis V, Cho SH, Goldberg S. Saphenous vein graft intervention: a review. J Invasive Cardiol. 2012 Feb;24(2):64-71. PMID 22294536
- [Background] Goldman S, Zadina K, Moritz T, Ovitt T, Sethi G, Copeland JG, Thottapurathu L, Krasnicka B, Ellis N, Anderson RJ, Henderson W; VA Cooperative Study Group #207/297/364. Long-term patency of saphenous vein and left internal mammary artery grafts after coronary artery bypass surgery: results from a Department of Veterans Affairs Cooperative Study. J Am Coll Cardiol. 2004 Dec 7;44(11):2149-56. doi: 10.1016/j.jacc.2004.08.064. PMID 15582312
- [Background] Lee MS, Park SJ, Kandzari DE, Kirtane AJ, Fearon WF, Brilakis ES, Vermeersch P, Kim YH, Waksman R, Mehilli J, Mauri L, Stone GW. Saphenous vein graft intervention. JACC Cardiovasc Interv. 2011 Aug;4(8):831-43. doi: 10.1016/j.jcin.2011.05.014. PMID 21851895
- [Background] Mehilli J, Pache J, Abdel-Wahab M, Schulz S, Byrne RA, Tiroch K, Hausleiter J, Seyfarth M, Ott I, Ibrahim T, Fusaro M, Laugwitz KL, Massberg S, Neumann FJ, Richardt G, Schomig A, Kastrati A; Is Drug-Eluting-Stenting Associated with Improved Results in Coronary Artery Bypass Grafts? (ISAR-CABG) Investigators. Drug-eluting versus bare-metal stents in saphenous vein graft lesions (ISAR-CABG): a randomised controlled superiority trial. Lancet. 2011 Sep 17;378(9796):1071-8. doi: 10.1016/S0140-6736(11)61255-5. Epub 2011 Aug 26. PMID 21872918
- [Background] Stone GW, Goldberg S, O'Shaughnessy C, Midei M, Siegel RM, Cristea E, Dangas G, Lansky AJ, Mehran R. 5-year follow-up of polytetrafluoroethylene-covered stents compared with bare-metal stents in aortocoronary saphenous vein grafts the randomized BARRICADE (barrier approach to restenosis: restrict intima to curtail adverse events) trial. JACC Cardiovasc Interv. 2011 Mar;4(3):300-9. doi: 10.1016/j.jcin.2010.11.013. PMID 21435608
- See also: link of the original (Swedish) project plan — https://www.researchweb.org/is/fourol/project/242381